CLINICAL TRIAL: NCT04279808
Title: Adequate Insertion Depth of Dilator During Central Venous Catheterization Through the Right Internal Jugular Vein
Brief Title: Adequate Insertion Depth of Dilator During Central Venous Catheterization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 10-2019-3
Record Dates: First submitted 2020-02-18; First posted 2020-02-21 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-02

CONDITIONS: Central Venous Catheterization

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- measured distance (Experimental): In the modified Seldinger's maneuver, after guide-wire insertion into the right internal jugular vein, "we will measure the distance between the skin puncture site and the outside of anterior wall of the jugular vein. Next, we will insert the dilator on the guidewire by the measured length."
  Interventions: Procedure: dilator depth
- conventional method (No Intervention): In the modified Seldinger's maneuver, after guide-wire insertion into the right internal jugular vein, "we will insert the dilator on the guidewire as commonly used method of the practitioners."

INTERVENTIONS:
Procedure: dilator depth — For soft tissue dilation just after guidewire insertion in central venous catheterization through the right internal jugular vein, investigators will measure the distance between the skin puncture site and outside of anterior wall of the vein with real-time ultrasonography in the measured depth group. Next, practitioner will insert the dilator by the measured length and continue to insert the central venous catheter. For the conventional group as a control group, practitioner will perform the central venous catheterization with a manner used routinely by the practitioner.
  Arms: measured distance

SUMMARY:
For safe central catheterization, clinicians must be aware of adequate dilator insertion depth not to directly dilate the venous wall. The purpose of the study is to find out adequate insertion depth of the dilator during central venous catheterization through the internal jugular vein with the aid of real-time ultrasonography.

DETAILED DESCRIPTION:
This randomized controlled trial is to compare the distance between the skin puncture site and the outside of anterior wall of the internal jugular vein measured by real-time ultrasonography with the conventional method which is routinely used in common clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* adult patients requiring central venous catheterization through the right internal jugular vein

Exclusion Criteria:

* suspicion for infection of the right neck site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
hematoma realted with the dilator | 1 Day (on the study day for each patient)
  hematoma from the vascular wall puncture by the dilator

SECONDARY OUTCOMES:
distance between skin puncture site and the outside of the anterior wall of the internal jugular vein | 1 Day (on the study day for each patient)
  distance between skin puncture site and the outside of the anterior wall of the internal jugular vein which will be measured by real-time ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Man Lee, M.D.,PhD, Principal Investigator — SMG-SNU Boramae Medical Center